CLINICAL TRIAL: NCT04155775
Title: Effects of a Platelet Transfusion Best Practices Alert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-47797
Record Dates: First submitted 2019-05-15; First posted 2019-11-07 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Thrombocytopenia
Keywords: Electronic Health Records; Best Practice Alerts
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Practice Alert (Experimental): Platelet transfusion orders for patients with a recent platelet count exceeding 50,000 per microliter (50k/uL) will trigger an alert in the electronic health record that displays current guidelines for platelet transfusion. The alert will allow providers to bypass the recommendation and continue with platelet ordering by selecting a clinical acknowledgement / exception to recommendation.Exclusions will be built into the alert to avoid triggering in operative or procedural settings, for neurosurgery providers, or patients on anti-platelet medications.
  Interventions: Other: Computer electronic health record alert (Best Practice Alert - BPA)
- No Best Practice Alert (No Intervention): For this group, no visible best practice alert will activate in the electronic health record for platelet transfusion orders and recent counts above 50k/uL.

INTERVENTIONS:
Other: Computer electronic health record alert (Best Practice Alert - BPA) — Upon ordering platelets in patients with recent platelet count >50,000, a pop-up within the electronic health system will recommend to not continue with transfuse product order and provide clinical exceptions to continue. Importantly, the alert does not trigger in operating areas, emergency medicine treatment areas, for certain specialties like neurosurgery or for massive transfusion orders.
  Arms: Best Practice Alert

SUMMARY:
This study is to determine the effectiveness of a computerized clinical decision support tool (Best Practice Alert - BPA) in reducing unnecessary platelet transfusions based on guidelines published by national transfusion societies such as the AABB (formerly American Association of Blood Banks).

DETAILED DESCRIPTION:
A computerized alert will be deployed through the electronic health record. The alert will trigger when a provider orders platelet transfusion above a threshold supported by current guidelines. The alert will provide information on current evidence and give the provider the option to cancel the order or proceed. The alert will not be triggered in procedural areas such as the operating room or as part of any emergency orders to prevent any delays to urgent patient care.

The proposed project will evaluate this alert by randomizing its implementation by patient chart. The investigators will observe the prevalence of this alert and its impact on ordering practices for the next 3 months. For patient charts randomized not to receive the intervention, the providers will not receive any alerts, but the analytics tool will record if the alert would have been triggered and the pertinent clinical information. After a period of three months, the investigators will review patient and provider information through analytics tools, assessing differences in platelet usage between the patients whose charts showed the alerts vs. those (control) patient charts not showing alerts.

ELIGIBILITY:
Inclusion Criteria:

* Recent platelet count >50k/uL
* Platelet transfusion ordered

Exclusion Criteria:

* Neurosurgery
* Procedure area (OR, catheterization lab, interventional radiology suite)
* Documented history of antiplatelet agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Platelet transfusions above threshold | Data will be initially reviewed before 6 months from start with anticipated completion 1 year from start
  Number of platelet transfusions occurring in patients with recent platelet counts above 50k/uL

SECONDARY OUTCOMES:
Total platelet transfusions | Data will be initially reviewed before 6 months from start with anticipated completion 1 year from start
  Total number of platelet transfusions occurring during study period.

CONTACTS AND LOCATIONS:
Overall Officials: Colin H Murphy, MD, Principal Investigator — Stanford University; Neil Shah, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Healthcare, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murphy C, Mou E, Pang E, Shieh L, Hom J, Shah N. A randomized study of a best practice alert for platelet transfusions. Vox Sang. 2022 Jan;117(1):87-93. doi: 10.1111/vox.13132. Epub 2021 Jun 3. PMID 34081800